CLINICAL TRIAL: NCT05907538
Title: Interoception in Patients With Medically Unexplained Symptoms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: TRACE labs Ziekenhuis Oost-Limburg (ZOL) (Unknown)
Responsible Party: Principal Investigator, Indra Ramakers, PhD researcher, Hasselt University
Other Study IDs: B1152021000014
Record Dates: First submitted 2023-05-24; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Fibromyalgia; Burnout, Psychological
Keywords: Fibromyalgia; Burnout; Interoception
MeSH Terms: conditions — Fibromyalgia; Burnout, Psychological

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with functional disorder (FD): Patients with fibromyalgia diagnosed using the ACR criteria (American College of Rheumatology, Wolfe et al., 2010; 2016) Patients with chronic fatigue syndrome diagnosed using the CDC criteria (Centers for Disease Control and Prevention; Fukuda et al., 1994)
  Interventions: Other: Interoceptive accuracy measurement; Other: Interoceptive sensibility measurement; Other: Interoceptive awareness measurement
- Patients with stress related syndromes (SRS): Patients with overstrain and burnout according to the multidisciplinary guidelines for overstrain and burnout in primary care from the Dutch Society of Occupational Medicine (NVAB, 2011)
  Interventions: Other: Interoceptive accuracy measurement; Other: Interoceptive sensibility measurement; Other: Interoceptive awareness measurement
- Healthy controls: Healthy controls will consist of people who experience few physical complaints in daily life. The healthy controls will thus be screened for inclusion using the CSD (Checklist for Symptoms in Daily life; Walentynowicz, et al., 2018). Only volunteers with a score of 75 or lower on this questionnaire will be included
  Interventions: Other: Interoceptive accuracy measurement; Other: Interoceptive sensibility measurement; Other: Interoceptive awareness measurement

INTERVENTIONS:
Other: Interoceptive accuracy measurement — Interoceptive accuracy will be measured using the Respiratory Occlusion Discrimination Task (ROD task; Van Den Houte et al., 2021). The ROD task measures how good subjects are at distinguishing the lengths of short (max 620 milliseconds) inspiratory occlusions (or respiratory interruptions).
Other: Interoceptive sensibility measurement — Interoceptive sensibility will be measured using two self-report questionnaires, the The Interoceptive Sensitivity and Attention Questionnaire (ISAQ; Bogaerts et al., 2022) and the the Three-domain Interoceptive Sensations Questionnaire (THISQ; Vlemincx et al., 2021)
Other: Interoceptive awareness measurement — Interoceptive awareness will be measures using a visual analogue scale (VAS)

SUMMARY:
The goal of this observational study is to learn about interoception in patients with stress related syndromes (overstrain, burnout; SRS) and functional disorder (fibromyalgia/ chronic fatigue syndrome; FD). The main questions it aims to answer are:

* Is there a significant difference in interoception between patients with SRS and healthy controls?
* Is there a significant difference in interoception between patients with FD and healthy controls?
* Is there a significant difference in interoception between patients with SRS and FD?

The participants will perform the respiratory occlusion discrimination task and have to fill out some questionnaires.

Researchers will compare healthy controls to see if there is a significant difference.

DETAILED DESCRIPTION:
About 40-49% of primary care patients report somatic symptoms that cannot be explained by any well-known organic disease. Typical examples are headache, dizziness, shortness of breath, fatigue, muscle aches, nausea, and gastrointestinal symptoms. These bodily symptoms can occur in the context of SRS such as overstrain and burnout, but also as clusters in a more chronic form, often referred to as FD, such as fibromyalgia or chronic fatigue syndrome.

Fibromyalgia is a chronic widespread pain condition characterized by point tenderness, fatigue, sleep disturbance, cognitive complaints, and increasing somatic complaints. In addition, chronic fatigue syndrome is a chronic condition characterized by severe fatigue, impairments in concentration and short-term memory, sleep disturbance, and musculoskeletal pain. Both are multi-faceted and challenging chronic conditions with considerable overlap in symptoms, causes and treatments. According to multidisciplinary guidelines, overstrain is characterized by the following symptoms: disturbed or restless sleep, irritability, not being able to stand commotion/ noise, emotional lability, feeling stressed or rushed, not being able to relax, difficulty concentrating and/or forgetfulness with a duration of 3 months. Burnout occurs when symptoms of overstrain persist for more than 6 months, and feelings of fatigue and exhaustion become prominent. The patient experiences significant limitations in professional and/or social functioning.

Interoception has been described in the literature as "the overall process of how the nervous system senses, integrates, stores and displays information about the state of the internal body". Theory suggests that interoception should be divided into three measurable constructs: interoceptive accuracy (objective accuracy in detecting internal bodily sensations), interoceptive sensitivity (the self-perceived tendency to be internally self-focused), and interoceptive awareness (metacognition about his/her own interoceptive accuracy).

The measurement will take place in the TRACE labs of Ziekenhuis Oost Limburg (ZOL). The informed consent will be signed before any data collection takes place. The experiment will take approximately 30 minutes. Participants will start with the interoceptive accuracy task using the Respiratory Occlusion Discrimination Task (ROD task). The ROD task measures how good subjects are at distinguishing the lengths of short (max 620 ms) inspiratory occlusions (or respiratory interruptions). Occlusions of these lengths are not aversive or unpleasant. One trial consists of two occlusions within one inspiration (inter-occlusion interval = 300 milliseconds), one occlusion being the reference occlusion (always 440 milliseconds) and one occlusion being the test occlusion (longer or shorter than 440 milliseconds), administered in random order. The participant is asked to indicate which of the two occlusions was longest. An adaptive staircase paradigm is used to determine the just noticeable difference in lengths of inspiratory occlusions. The length of the task depends on the performance of the subject, but is on average 56 trials (= 15 minutes). After the experiment, another short side experiment of 16 trials will be conducted in which the participant should indicate how confident they were in their response on a Visual Analogue scale (VAS), in order to estimate interoceptive awareness. In the meantime, participants will be also asked to complete a questionnaire bundle at home (online), which takes approximately 45 minutes to complete.

The power calculations resulted in a total of 28 persons per group. Therefore the investigators plan to recruit a total of 84 people.

Primary outcomes are interoceptive accuracy, interoceptive sensibility, and interoceptive awareness. Secondary outcome measures are psychological variables measured using questionnaires.

Descriptive statistics will be used to display baseline group characteristics. To evaluate between-group differences (i.e. the difference between patients with FD,SRS and healthy controls regarding interoception and psychological variables) one-way ANOVA's will be used.

ELIGIBILITY:
Eligibility Criteria patients with FD (fibromyalgia and/or chronic fatigue syndrome)

Inclusion Criteria:

* patients with fibromyalgia should be diagnosed by using the ACR criteria (American College of Rheumatology, Wolfe et al., 2010; Wolfe et al., 2016). patients with chronic fatigue syndrome should be diagnosed by using the CDC criteria (Centers for Disease Control and Prevention; Fukuda et al., 1994).

Exclusion Criteria:

* Younger than 18 or older than 65
* Pregnancy
* Primary depressive episode, anxiety disorder, eating disorder, substance abuse, neurocognitive, or psychotic episode diagnosed with DSM-V (Diagnostic and Statistical Manual of Mental Disorders; MINI-s; Overbeek et al., 1999).
* Presence of a chronic organic disorder (One speaks of a chronic organic disorder if it is present for a period of at least 3 months. Examples include: Epilepsy, Heart Disease, Rheumatism, Asthma, Diabetes, etc.) or acute organic condition (fever, flu, etc.)
* BMI > 30

Eligibility Criteria patients with SRS (overstrain or burnout)

Inclusion Criteria:

- patients with overstrain or burnout should be diagnosed according to the multidisciplinary guidelines for overstrain and burnout for first-line professionals from the Dutch Society of Occupational Medicine (NVAB, 2011)

Exclusion Criteria:

* Younger than 18 or older than 65
* Pregnancy
* Primary depressive episode, anxiety disorder, eating disorder, substance abuse, neurocognitive, or psychotic episode diagnosed with DSM-V (MINI-s; Overbeek et al., 1999).
* Presence of a chronic organic disorder (One speaks of a chronic organic disorder if it is present for a period of at least 3 months. Examples include: Epilepsy, Heart Disease, Rheumatism, Asthma, Diabetes, etc.) or acute organic condition (fever, flu, etc.)
* BMI > 30

Eligibility Criteria healthy controls

Inclusion Criteria:

Healthy controls will be selected so that there is an equal ratio between patients and healthy controls for

* Age group (per 5 years)
* Gender (including X)
* Educational attainment
* BMI

all participants need a score < 75 on the CSD (Walentynowicz, et al., 2018)

Exclusion Criteria:

* Younger than 18 or older than 65
* Pregnancy
* Presence of a depressive episode, anxiety disorder, eating disorder, substance abuse, neurocognitive, or psychotic disorder diagnosed with DSM-V (MINI-s; Overbeek et al., 1999).
* Presence of a chronic organic disorder (One speaks of a chronic organic disorder if it is present for a period of at least 3 months. Examples are: epilepsy, heart disease, rheumatism, asthma, diabetes, etc.) or acute organic disorder (fever, flu, etc.)
* BMI > 30
* Persistent physical symptoms (e.g., hyperventilation symptoms, prolonged COVID, chronic pain or fatigue, chronic tinnitus, etc.)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients with fibromyalgia diagnosed according to the ACR criteria (Wolfe et al., 2010; 2016) are eligible to participate, all patients with chronic fatigue syndrome diagnosed according to the CDC criteria (Fukuda et al., 1994), and all patients with overstrain or burnout diagnosed according to the multidisciplinary guidelines for overstrain and burnout for first-line professionals from the Dutch Society of Occupational Medicine (NVAB, 2011) are eligible to participate
Sampling Method: Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Interoceptive accuracy | 20 minutes
  Respiratory occlusion discrimination task (ROD task; Van Den Houte et al., 2021)
Interoceptive sensibility | 5 minutes
  Interoceptive Sensitivity and Attention Questionnaire (ISAQ; Bogaerts et al., 2022)
Interoceptive sensibility | 5 minutes
  THree-domain Interoceptive Sensations Questionnaire (THISQ; Vlemincx et al., 2021)
Interoceptive awareness | 5 minutes
  Visual analogue scale (0-100). A score of 0 indicates that participants are not certain at all of their answer, a score of 100 indicates that participants are entirely certain of their answer

SECONDARY OUTCOMES:
Psychological variables | 5 minutes
  Checklist for Symptoms in Daily Life (CSD; Walentynowicz et al., 2018)
Psychological variables | 5 minutes
  Positive and Negative Affect Scale (PANAS; Watson et al., 1988)
Psychological variables | 5 minutes
  Tellegen Absorption Scale (TAS; Tellegen & Atkinson, 1974)
Psychological variables | 10 minutes
  Traumatic Experiences Checklist (TEC; Nijenhuis et al., 2002)
Psychological variables | 5 minutes
  Toronto Alexithymia Scale (TAS-20; Bagby et al., 1994)
Psychological variables | 5 minutes
  Need for Controllability and Predictability Questionnaire (NCP-q; Ramakers et al., manuscript in preparation)
Psychological variables | 5 minutes
  Frost Multidimensional Perfectionism Scale (FMPS; Frost et al., 1990)
Psychological variables | 5 minutes
  Acceptance and Action Questionnaire-II (AAQ-II; Bond et al., 2011)

CONTACTS AND LOCATIONS:
Overall Officials: Katleen Bogaerts, PhD, Principal Investigator — Hasselt University
Locations (2):
- Belgium (2):
  - Hasselt University, Diepenbeek, Limburg
  - TRACE labs Ziekenhuis Oost-Limburg (ZOL), Lanaken

REFERENCES:
- [Background] Haller H, Cramer H, Lauche R, Dobos G. Somatoform disorders and medically unexplained symptoms in primary care. Dtsch Arztebl Int. 2015 Apr 17;112(16):279-87. doi: 10.3238/arztebl.2015.0279. PMID 25939319
- [Background] Barsky AJ, Borus JF. Functional somatic syndromes. Ann Intern Med. 1999 Jun 1;130(11):910-21. doi: 10.7326/0003-4819-130-11-199906010-00016. PMID 10375340
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Katz RS, Mease P, Russell AS, Russell IJ, Winfield JB, Yunus MB. The American College of Rheumatology preliminary diagnostic criteria for fibromyalgia and measurement of symptom severity. Arthritis Care Res (Hoboken). 2010 May;62(5):600-10. doi: 10.1002/acr.20140. PMID 20461783
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RL, Mease PJ, Russell AS, Russell IJ, Walitt B. 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria. Semin Arthritis Rheum. 2016 Dec;46(3):319-329. doi: 10.1016/j.semarthrit.2016.08.012. Epub 2016 Aug 30. PMID 27916278
- [Background] Walentynowicz, M., Witthöft, M., Raes, F., Van Diest, I., & Van den Bergh, O. (2018). Sensory and affective components of symptom perception: a psychometric approach. Journal of Experimental Psychopathology, 9(2), 1-13. Doi: 10.5127/jep.059716
- [Background] Courtois I, Cools F, Calsius J. Effectiveness of body awareness interventions in fibromyalgia and chronic fatigue syndrome: a systematic review and meta-analysis. J Bodyw Mov Ther. 2015 Jan;19(1):35-56. doi: 10.1016/j.jbmt.2014.04.003. Epub 2014 Apr 18. PMID 25603742
- [Background] NVAB. (2011). Eén lijn in de eerste lijn bij overspanning en burnout: Multidisciplinaire richtlijn overspanning en burnout voor eerstelijns professionals. Geraadpleegd van https://nvab-online.nl/sites/default/files/bestanden-webpaginas/MDRL_Overspanning-Burnout.pdf
- [Background] Terluin, B., Van der Klink, J., Schaufeli, W. (2005). Stressgerelateerde klachten: spanningsklachten, overspanning en burnout. In J. Van der Klink, B. Terluin B (Reds), Psychische problemen en werk. Handboek voor een activerende begeleiding door huisarts en bedrijfsarts (p. 259-290). Houten: Bohn Stafleu Van Loghum.
- [Background] van der Klink JJ, van Dijk FJ. Dutch practice guidelines for managing adjustment disorders in occupational and primary health care. Scand J Work Environ Health. 2003 Dec;29(6):478-87. doi: 10.5271/sjweh.756. PMID 14712856
- [Background] Khalsa SS, Adolphs R, Cameron OG, Critchley HD, Davenport PW, Feinstein JS, Feusner JD, Garfinkel SN, Lane RD, Mehling WE, Meuret AE, Nemeroff CB, Oppenheimer S, Petzschner FH, Pollatos O, Rhudy JL, Schramm LP, Simmons WK, Stein MB, Stephan KE, Van den Bergh O, Van Diest I, von Leupoldt A, Paulus MP; Interoception Summit 2016 participants. Interoception and Mental Health: A Roadmap. Biol Psychiatry Cogn Neurosci Neuroimaging. 2018 Jun;3(6):501-513. doi: 10.1016/j.bpsc.2017.12.004. Epub 2017 Dec 28. PMID 29884281
- [Background] Garfinkel SN, Seth AK, Barrett AB, Suzuki K, Critchley HD. Knowing your own heart: distinguishing interoceptive accuracy from interoceptive awareness. Biol Psychol. 2015 Jan;104:65-74. doi: 10.1016/j.biopsycho.2014.11.004. Epub 2014 Nov 20. PMID 25451381
- [Background] Van Den Houte M, Vlemincx E, Franssen M, Van Diest I, Van Oudenhove L, Luminet O. The respiratory occlusion discrimination task: A new paradigm to measure respiratory interoceptive accuracy. Psychophysiology. 2021 Apr;58(4):e13760. doi: 10.1111/psyp.13760. Epub 2021 Jan 12. PMID 33438245
- [Background] Fukuda K, Straus SE, Hickie I, Sharpe MC, Dobbins JG, Komaroff A. The chronic fatigue syndrome: a comprehensive approach to its definition and study. International Chronic Fatigue Syndrome Study Group. Ann Intern Med. 1994 Dec 15;121(12):953-9. doi: 10.7326/0003-4819-121-12-199412150-00009. PMID 7978722
- [Background] Bogaerts K, Walentynowicz M, Van Den Houte M, Constantinou E, Van den Bergh O. The Interoceptive Sensitivity and Attention Questionnaire: Evaluating Aspects of Self-Reported Interoception in Patients With Persistent Somatic Symptoms, Stress-Related Syndromes, and Healthy Controls. Psychosom Med. 2022 Feb-Mar 01;84(2):251-260. doi: 10.1097/PSY.0000000000001038. PMID 34840287
- [Background] Vlemincx E, Walentynowicz M, Zamariola G, Van Oudenhove L, Luminet O. A novel self-report scale of interoception: the three-domain interoceptive sensations questionnaire (THISQ). Psychol Health. 2023 Sep-Oct;38(9):1234-1253. doi: 10.1080/08870446.2021.2009479. Epub 2021 Dec 7. PMID 34875958
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Background] Nijenhuis, E. R. S., van der Hart, O., & Kruger, K. (2002). The psychometric characteristics of the Traumatic Experiernce Checklist (TEC): First findings among psychiatric outpatients. Clinical Psychology & Psychotherapy, 9(3). 200-210. DOI: 10.1002/cpp.332
- [Background] Bagby RM, Parker JD, Taylor GJ. The twenty-item Toronto Alexithymia Scale--I. Item selection and cross-validation of the factor structure. J Psychosom Res. 1994 Jan;38(1):23-32. doi: 10.1016/0022-3999(94)90005-1. PMID 8126686
- [Background] Bond FW, Hayes SC, Baer RA, Carpenter KM, Guenole N, Orcutt HK, Waltz T, Zettle RD. Preliminary psychometric properties of the Acceptance and Action Questionnaire-II: a revised measure of psychological inflexibility and experiential avoidance. Behav Ther. 2011 Dec;42(4):676-88. doi: 10.1016/j.beth.2011.03.007. Epub 2011 May 25. PMID 22035996
- [Background] Frost, R. O., Marten, P., Lahart, C., & Rosenblate, R. (1990). The dimensions of perfectionism. Cognitive Therapy and Research, 14(5), 449-468. https://doi.org/10.1007/BF01172967
- [Background] Tellegen A, Atkinson G. Openness to absorbing and self-altering experiences ("absorption"), a trait related to hypnotic susceptibility. J Abnorm Psychol. 1974 Jun;83(3):268-77. doi: 10.1037/h0036681. No abstract available. PMID 4844914
- [Background] Overbeek, T., Schrueurs, K., & Griez, E. (1999). MINI-the international neuropsychiatric interview. Dutch version 5.0.0 DSM-IV. Maastricht (Netherlands): University of Maastricht.
- [Background] Ramakers I, Fonteyne R, Walentynowicz M, Oudenhove LV, Houte MVD, Bogaerts K. The Need for Controllability and Predictability questionnaire (NCP-q): psychometric properties and preliminary findings in a clinical sample. Health Psychol Rep. 2025 Jan 24;13(2):201-214. doi: 10.5114/hpr/195733. eCollection 2025. PMID 40487476